CLINICAL TRIAL: NCT03723603
Title: A Case Series Evaluating a Fibrillar Collagen Powder Dressing to Treat Chronic, Stalled Lower-extremity Wounds
Brief Title: An Evaluation of a Collagen Dressing to Treat Chronic, Stalled Lower-extremity Wounds
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to a re-prioritization of ongoing studies.
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MED-2018-DIV71-018
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Results first posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-02

CONDITIONS: Wound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Fibrillar Collagen Powder Dressing (Experimental)
  Interventions: Device: Fibrillar collagen powder dressing

INTERVENTIONS:
Device: Fibrillar collagen powder dressing — A powder-like fibrillar collagen microsponge composed of Type I porcine dermis collagen. The dressing is a currently marketed, cleared device in the United States, indicated for the management of full and partial thickness wounds: pressure ulcers, diabetic ulcers, caused by mixed vascular origin, venous ulcers, and several other wound types.

SUMMARY:
Patients who meet the inclusion criteria will be provided with fibrillar collagen powder dressing. The powder dressing will be used in accordance with its label. After cleansing the wound by the clinical site staff, the powder is placed directly on the wound, and then the wound will be covered with an appropriate moisture retentive secondary dressing. Patients will visit the clinic twice a week to have the powder re-applied. Wound evaluations will take place once a week at the outpatient clinic, with the intervention lasting up to twelve weeks. Concurrent standard of care, such as compression for venous ulcers, will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Has one of the following types of wounds below the knee: diabetic ulcers, pressure ulcers, venous ulcers, ulcers of mixed-vascular origin, traumatic wounds, or post-surgical wounds
* Wound has been present for at least four weeks
* Wound is free of necrotic tissue or debridement practices will take place prior to initial visit in order to remove necrotic tissue
* Wound has failed at least one wound care treatment
* Wound size is between 1 and 100 square centimeters
* Patient has adequate circulation as demonstrated by biphasic or triphasic Doppler waveform, measured within three months prior to study enrollment. If monophasic on exam, then non-invasive tests must display Ankle Brachial Index greater than 0.8 and no worse than mild disease on segmental pressures.
* Wound is confirmed as being free of infection and absence of osteomyelitis

Exclusion Criteria:

* Pregnant, planning to become pregnant during the study timeframe, or breast feeding
* Unable or unwilling to receive porcine collagen
* Wound is infected or presence of osteomyelitis
* Allergy or sensitivity to collagen
* Inability, in the opinion of the Investigator to follow protocol requirements, attend follow up visits in a timely manner, or otherwise comply with the requirements of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Windy Cole, Principal Investigator — Cleveland Foot and Ankle Clinic
Locations (1):
- Cleveland Foot and Ankle Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fibrillar Collagen Powder Dressing
Started | 8
Completed | 5
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Study terminated prematurely due to re-prioritization of study efforts. Data not assessed.
Arm/Group | Fibrillar Collagen Powder Dressing
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race/Ethnicity, Customized
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Change in Wound Size Over Twelve Week Period
Time Frame: Baseline to 84 days
Population: Study terminated prematurely due to re-prioritization of study efforts. Data not assessed.
Arm/Group | Fibrillar Collagen Powder Dressing
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in Bates-Jensen Wound Assessment Tool
Description: The Bates-Jensen Wound Assessment tool score will be used to assess the wound's status throughout the study. The Bates-Jensen Wound Assessment tool measures wound status. The wound size score ranges from 0 to 5. The wound depth score ranges from 0 to 5. The wound edge score ranges from 0 to 5. The wound undermining score ranges from 0 to 5. The necrotic tissue type score ranges from 1 to 5. The necrotic tissue amount ranges from 1 to 5. The exudate type score ranges from 1 to 5. The exudate amount score ranges from 1 to 5. The skin color surrounding wound score ranges from 1 to 5. The peripheral tissue edema score ranges from 1 to 5. The peripheral tissue induration score score ranges from 1 to 5. The granulation tissue score ranges from 1 to 5. The epithelialization score ranges from 1 to 5. The total score from these sub-scores added together is used as the total BWAT score. For all sub-score values, a value of 0 or 1 is a better outcome.
Time Frame: Baseline to 84 days
Population: Study terminated prematurely due to re-prioritization of study efforts. Data not assessed.
Arm/Group | Fibrillar Collagen Powder Dressing
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Reported Pain Level
Description: The pain score will be recorded with a verbal numeric pain rating scale from 0-10.
Time Frame: Baseline to 84 days
Population: Study terminated prematurely due to re-prioritization of study efforts. Data not assessed.
Arm/Group | Fibrillar Collagen Powder Dressing
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline to 12 weeks
Description: Study terminated prematurely due to re-prioritization of study efforts. Serious Adverse Events were assessed and reported. Other non serious adverse events were not assessed.
Arm/Group | Fibrillar Collagen Powder Dressing
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 3/3
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fibrillar Collagen Powder Dressing (N=3)
Death (Cardiac disorders) | 1
Infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-21): https://cdn.clinicaltrials.gov/large-docs/03/NCT03723603/Prot_SAP_000.pdf